CLINICAL TRIAL: NCT03696303
Title: Determination of the Utility of Pfizer's Pneumococcal Urine Antigen Test in Children 5 Years of Age or Younger With Community Acquired Pneumonia in Guatemala
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18-0737
Record Dates: First submitted 2018-10-01; First posted 2018-10-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Community-acquired Pneumonia; Streptococcus Pneumoniae Infection
Keywords: Streptococcus pneumoniae; Pneumonia; Community-acquired; Pediatric; Urine antigen
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumococcal Infections; Pneumonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine Blood Nasopharyngeal swab samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cases: Suspected community-acquired bacterial pneumonia
  Interventions: Other: Urinary antigen detection assay
- Controls: Healthy children, age-matched to enrolled cases
  Interventions: Other: Urinary antigen detection assay
- Controls with URI: Children 5 years of age or younger with upper respiratory infection (URI) (controls with URI)
  Interventions: Other: Urinary antigen detection assay

INTERVENTIONS:
Other: Urinary antigen detection assay — Screening for Ag level in S. pneumoniae urinary antigen detection assay.

SUMMARY:
This prospective case-control study aims to evaluate the utility and establish laboratory thresholds for a multi-serotype urine antigen test for the diagnosis of pneumococcal community acquired pneumonia in children 5 years of age or younger in Guatemala.

ELIGIBILITY:
CASES:

Inclusion Criteria:

* Age older than 1 month (31 days) and up to 71 months and 28 days.
* Diagnosis of radiologically confirmed pneumonia per WHO criteria in the ED or hospital within 48 hours of hospital admission
* Signed informed consent by parents or legal guardian to participate in the study

Exclusion Criteria:

* Known immunodeficiency
* Major congenital malformation (e.g., hemodynamically compromised congenital heart malformation or any malformation leading to recurrent pneumonia) or serious chronic disorder
* Significant neurological disorder
* Hospitalization within the previous 30 days for pneumonia or respiratory infection
* Use of parenteral antibiotics for current illness (leading to diagnosis of pneumonia)
* Transferred to the study hospital after already being hospitalized at a different location for ≥ 48 hours

CONTROLS:

Inclusion Criteria:

* Age 1 to 71 months and signed informed consent by parents or legal guardian

Exclusion Criteria:

* Known immunodeficiency
* Major congenital malformation (e.g., hemodynamically compromised congenital heart malformation or any malformation leading to recurrent pneumonia) or serious chronic disorder
* Significant neurological disorder
* Fever or suspicion of community-acquired pneumonia or other respiratory infectious disease (symptoms of cough, congestion, tachypnea, indrawing, etc.)
* Hospitalization within the previous 30 days for pneumonia or respiratory infection

Ages: 31 Days to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children 5 years of age or younger with either community-acquired pneumonia (cases) or health children (controls).
Sampling Method: Non-Probability Sample
Enrollment: 959 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Urinary antigen detection cut-points for invasive S. pneumoniae disease | Within 48 hours
  To determine Cut-Points to discriminate a positive or negative urine antigen test that differentiates invasive disease versus the carriage state

SECONDARY OUTCOMES:
Detection of S. pneumoniae serotypes using Urinary antigen detection assay | Within 48 hours
  To determine the sensitivity and specificity of the Luminex xMPA pneumococcal UAD in the identification of S. pneumoniae serotypes (PCV13 serotypes) in children with radiologically confirmed CAP

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Asturias, MD, Principal Investigator — University of Colorado, Denver
Locations (3):
- Guatemala (3):
  - Hospital Regional Cuilapa, Cuilapa, Santa Rosa Department
  - Hospital General IGSS, Guatemala City
  - Hospital Roosevelt, Guatemala City

IPD SHARING:
Plan to Share IPD: No